CLINICAL TRIAL: NCT04361071
Title: Clinical Study of Stent Versus Direct Atherectomy to Treat Iliac Artery Occlusive Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XuanwuHvas
Record Dates: First submitted 2017-12-27; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2019-08

CONDITIONS: Iliac Artery Occlusion
Keywords: stent; atherectomy; iliac Artery
MeSH Terms: interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Stent (Active Comparator): Stent group
  Interventions: Device: stent
- Atherectomy (Active Comparator): Atherectomy group
  Interventions: Device: plaque excision system

INTERVENTIONS:
Device: stent — stent
  Arms: Stent
Device: plaque excision system — plaque excision system
  Arms: Atherectomy

SUMMARY:
This is a randomized study comparing stent and plaque excision systems in treatment of Iliac artery occlusive disease.

DETAILED DESCRIPTION:
This is a randomized study comparing stent and plaque excision systems in treatment of Iliac artery occlusive disease

ELIGIBILITY:
Inclusion Criteria:

1. The patients have non thrombotic arteriosclerosis obliterans of the common iliac or external iliac arteries
2. Clinical diagnosis of stenosis or occlusive disease
3. The patients have unobstructed distal outflow tract
4. Receiving surgical treatment at the same time

Exclusion Criteria:

1. The patients who have previously implanted stent(s) or stent graft(s) in target leg
2. Life expectancy less than 12 months
3. Has any planned surgical or endovascular intervention of target vessel 30 days before or after index procedure
4. Thrombophlebitis, uremia, or deep venous thrombus, within past 30 days
5. Receiving dialysis or immunosuppressant therapy
6. Recent stroke within past 90 days
7. Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix®) or ticlopidine (Ticlid®), heparin, Nitinol (nickel titanium), contrast agent, that cannot be medically managed
8. Tissue loss due to ischemic disease (Rutherford/Becker category 5 or 6)
9. Serum creatinine level >/= 2.5 mg/dl at time of screening visit
10. Known or suspected active infection at the time of the procedure
11. Bleeding diathesis
12. Patient is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol.
13. Patients are known to be pregnant, incarcerated, mentally incompetent, and/or alcohol or drug abuser.
14. Patients are currently participating in any other investigational drug or medical device study that has not completed primary endpoint(s) evaluation or clinically interferes with the endpoints from this study or future participation in such studies prior to the completion of this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
12-month Primary Patency Rate | 12 months
  Primary patency is defined as no significant reduction of flow detectable by Duplex ultrasound through the index lesion and no further clinically driven target vessel revascularization performed in the interim. Significant reduction of flow is binary restenosis defined as the diameter stenosis >50% with a peak systolic velocity ratio >2.4 as measured by Duplex ultrasound.
12-month Limb Salvage Rate | 12 months
  Limb Salvage is defined as the freedom from secondary major amputation

SECONDARY OUTCOMES:
Index Limb Ischemia at 6-month Follow up | 6 months
  Index Limb Ischemia is defined by Rutherford/Becker Classification categories 3 through 6.
Index Limb Ischemia at 12-month Follow up | 12 months
  Index Limb Ischemia is defined by Rutherford/Becker Classification categories 3 through 6.
Major Adverse Events at 12-month Post Procedure | 12 months
  Major adverse events included death, index limb ischemia, index limb amputation, clinically driven target lesion revascularization , and significant embolic events, which were defined as causing end-organ damage.

CONTACTS AND LOCATIONS:
Locations (1):
- Yongquan Gu, Beijing, Beijing Municipality, China